CLINICAL TRIAL: NCT01757028
Title: Risk Factors for Severe Morbidity and Mortality in Mothers and Neonates
Acronym: KIPMAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: B9RPET0
Record Dates: First submitted 2012-11-28; First posted 2012-12-28 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Maternal and Newborn Health
Keywords: Maternal and newborn health; Africa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cord blood Maternal blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Improving maternal and infant mortality are key priorities in Kenya and internationally. This study aims to establish a hospital-based surveillance system for pregnant women so that the contribution of risk factors (HIV and other infections, maternal nutrition, sepsis, malaria and anaemia) to maternal and infant morbidity and mortality can be accurately assessed. All mothers who are admitted to Kilifi District Hospital will be invited to enrol in the study. Routine clinical data from maternal admissions for delivery will be systematically collected using a standardised admissions procedure. Analysis will be carried out for the risk factor effects of HIV, maternal nutrition, malaria infection, bacterial infection, and anaemia on maternal and infant outcomes after adjusting for other factors (mode of delivery, age, and parity etc). Subsequent morbidity and survival of mothers and infants, and the later consequences to children's health will be monitored through the Kilifi epi-DSS. Samples for research purposes will be collected for detailed future studies of particular pathogens and risk factors, such as malaria parasite strain, bacterial species and HIV-induced immunological impairment. This will be the first prospective study in sub-Saharan Africa (sSA) to assess the effect of these risk factors on both maternal and infant health together, and that considers both short and long term outcomes. Information generated by the study will be used by the maternity department in a rolling audit that will help improve care. The study will therefore improve care of new mothers and infants attending the Kilifi District Hospital as well as informing health planning so that future interventions for maternal and child health are targeted more effectively.

ELIGIBILITY:
Inclusion Criteria:

* All mothers admitted for delivery at Kilifi District Hospital (KDH), Kilifi, Kenya

Exclusion Criteria:

* Consent refusal

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All mothers admitted for delivery at Kilifi District Hospital (KDH), Kilifi, Kenya
Sampling Method: Probability Sample
Enrollment: 4600 (Estimated)
Dates: Start 2010-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Maternal mortality | At delivery and follow up through DHS to 42 days
  Determine the effects of risk factors and obstetric events on maternal deaths (to 42 days).
Perinatal mortality | To 7 days post delivery
  Determine the effects of risk factors and obstetric events on perinatal mortality (stillbirth and deaths to 7 days of life); infant mortality to 60 days

SECONDARY OUTCOMES:
Maternal and Newborn long term survival | ongoing
  Follow up to 2 years after delivery
Maternal morbidity | During admission (about 3 days)
  Life threatening events and maternal conditions at delivery
Neonatal morbidity | During admission (approx 2 weeks if admitted)
  Neonatal morbidity in terms of admission to the paediatric ward (and diagnosis).

CONTACTS AND LOCATIONS:
Locations (1):
- Kilifi District Hospital, Kilifi, Coast, Kenya